CLINICAL TRIAL: NCT04193137
Title: Comparison of Saline Infusion Test, Captopril Challenge Test, and Oral Sodium Loading Test in the Diagnosis of Primary Aldosteronism
Brief Title: Comparison of Three Confirmatory Tests in the Diagnosis of Primary Aldosteronism
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qifu Li, Primary Investigator, Chongqing Medical University
Other Study IDs: OSL-study 2019
Record Dates: First submitted 2019-12-08; First posted 2019-12-10 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Primary Aldosteronism
Keywords: primary aldosteronism,; oral sodium loading test; captopril challenge test,; Saline infusion test
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma and complete blood cell. 24-h urine, etc
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Aldosteronism(PA): plasma aldosterone /renin ratio (ARR)>10 pg/μIU and plasma aldosterone concentration(PAC) post-FST≥60pg/ml；or PAC>200 pg/ml，plasma renin concentration(PRC)<2.5μIU/ml，with hypokalemia
  Interventions: Diagnostic Test: Oral sodium loading test,Seated saline infusion test and Captopril challenge test
- non Primary Aldosteronism: ARR<10 pg/μIU or ARR>10 pg/μIU and PAC post FST<60pg/ml
  Interventions: Diagnostic Test: Oral sodium loading test,Seated saline infusion test and Captopril challenge test

INTERVENTIONS:
Diagnostic Test: Oral sodium loading test,Seated saline infusion test and Captopril challenge test — Oral sodium loading test : Patients received 6g oral sodium every day for 3 days.
  Seated saline infusion test: All participants received the infusion of 2 liters of 0.9% saline over 4 h in seated posture.
  Captopril challenge test: Patients received 50 mg captopril orally at 8-9 a.m. after sitting or standing for at least 2 h. Blood samples were drawn at time zero and 2 h after the challenge.

SUMMARY:
To compare the diagnostic value of three confirmatory tests for primary aldosteronism.

DETAILED DESCRIPTION:
This is a prospective study involving 240 hypertensive patients who underwent primary aldosteronism screening. Every patient will undertake four confirmatory tests to compare the diagnostic accuracy of the oral sodium loading test with captopril challenge testing (CCT) and Seated saline infusion test(SSST)using the fludrocortisone suppression testing (FST) as the reference standard, and to investigate the optimal cutoff of oral sodium loading test

ELIGIBILITY:
Inclusion Criteria:

1. hypertensive patients with ARR≥10(pg/ml)(uIU/ml)
2. hypertensive patients with ARR<10(pg/ml)(uIU/ml) but suspicious of PA clinically

Exclusion Criteria:

1. Pregnancy or lactation;
2. Child-bearing women refuse to take effective contraceptive measures;
3. History of malignant tumor;
4. Patients with cardiovascular and cerebrovascular diseases (eg. myocardial infarction, acute heart failure, stroke), in the past 3 months
5. NYHA III (New York Heart Association)and above
6. Hypohepatia
7. Chronic kidney disease with an estimated Glomerular Filtration Rate <30ml/min/1.73 m²
8. Severe arrhythmia by ECG or severe heart disease by cardiac ultrasound
9. Patients who are unwilling to participate in and complete this study and refuses to sign the informed consent form for this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hypertensive patients being suspicious of PA in a single tertiary hospital center
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of oral sodium loading test, captopril challenge test and saline infusion test | 9 days
  sensitivity, specificity and area under curve (AUC)

SECONDARY OUTCOMES:
the optimal cutoff value of urine aldosterone in oral sodium test | 3 days
  urine aldosterone

CONTACTS AND LOCATIONS:
Overall Officials: Qifu Li, PhD, Study Chair — the Chongqing Primary Aldosteronism Study (CONPASS) Group
Locations (1):
- Qifu Li, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Result] Young WF Jr. Diagnosis and treatment of primary aldosteronism: practical clinical perspectives. J Intern Med. 2019 Feb;285(2):126-148. doi: 10.1111/joim.12831. Epub 2018 Sep 25. PMID 30255616
- [Result] Wu S, Yang J, Hu J, Song Y, He W, Yang S, Luo R, Li Q. Confirmatory tests for the diagnosis of primary aldosteronism: A systematic review and meta-analysis. Clin Endocrinol (Oxf). 2019 May;90(5):641-648. doi: 10.1111/cen.13943. Epub 2019 Feb 26. PMID 30721529
- [Result] Mulatero P, Milan A, Fallo F, Regolisti G, Pizzolo F, Fardella C, Mosso L, Marafetti L, Veglio F, Maccario M. Comparison of confirmatory tests for the diagnosis of primary aldosteronism. J Clin Endocrinol Metab. 2006 Jul;91(7):2618-23. doi: 10.1210/jc.2006-0078. Epub 2006 May 2. PMID 16670162
- [Result] Nishikawa T, Omura M, Satoh F, Shibata H, Takahashi K, Tamura N, Tanabe A; Task Force Committee on Primary Aldosteronism, The Japan Endocrine Society. Guidelines for the diagnosis and treatment of primary aldosteronism--the Japan Endocrine Society 2009. Endocr J. 2011;58(9):711-21. doi: 10.1507/endocrj.ej11-0133. Epub 2011 Aug 9. PMID 21828936
- [Result] Mulatero P, Monticone S, Burrello J, Veglio F, Williams TA, Funder J. Guidelines for primary aldosteronism: uptake by primary care physicians in Europe. J Hypertens. 2016 Nov;34(11):2253-7. doi: 10.1097/HJH.0000000000001088. PMID 27607462